CLINICAL TRIAL: NCT01585181
Title: A Phase 1 Randomized, Double-Blind Placebo Controlled Study to Evaluate the Safety and Immunogenicity of the LIve Oral Cholera Vaccine Candidate PXVX0200 Vibrio Cholerae Serotype 01 Inaba CVD 103-HgR Vaccine Strain
Brief Title: Safety and Immunogenicity of the Live Oral Cholera Vaccine Candidate PXVX0200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PXVX-VC-0200-002
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cholera
Keywords: Vaccine, Bacterial disease condition, Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- PXVX0200 (Experimental)
  Interventions: Biological: PXVX0200

INTERVENTIONS:
Biological: PXVX0200 — Single dose; liquid suspension after reconstitution with buffer; 2x108 to 2x109 CFU in a liquid suspension
  Arms: PXVX0200
Biological: Placebo — Approx 2 grams of lactose reconstituted in water
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and immunogenicity of a single dose of the PXVX0200 live cholera vaccine versus placebo in volunteers (Vaccinees) and whether PXVX0200, which is a live attenuated bacteria, can be transmitted to other adults living in the same household.

DETAILED DESCRIPTION:
Approximately 60 subjects and up to 120 household contacts will be enrolled in the United States. Vaccinees will be randomly assigned to receive either PXVX0200 or placebo in a 5:1 ratio and will be followed for 180 days postdose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men or women, age 18 to 50 years (inclusive) without significant medical history, physical or clinical lab abnormalities (as per protocol defined ranges)
* Women of childbearing potential must have negative urine pregnancy test and must be willing to use adequate birth control for 2 months following vaccination and have additional pregnancy tests as indicated
* Vaccinees must live alone or have no more than two household contacts willing to sign informed consent and participate in the study
* Household contacts must be healthy (based on medical history) men or women aged 18-65 years (inclusive)

Exclusion Criteria:

* Healthcare workers who have direct contact with patients who are immunodeficient, are HIV-positive, have unstable medical condition or are under the age of 18
* Childcare workers who have direct contact with children who are 2 years of age or younger or those employed in the food service industry
* Resides with HHCs who are under the age of 18 or over the age of 65
* Has abnormal stool pattern defined as fewer than 3 stools per week or more than 2 stools per day in past 6 months
* Has known allergy to, or known medical condition that precludes the use of both tetracycline or ciprofloxacin
* Previously received a licensed or investigational cholera vaccine
* Has history of cholera or enterotoxigenic E. coli infection (natural infection or experimental challenge)
* Travel to a cholera-endemic area and experienced symptoms consistent with traveler's diarrhea in the previous 5 years
* Received or plans to receive any other licensed vaccines from 14 days prior to the study vaccination until Day 28
* Received or plans to receive antibiotics (other than protocol-specified) or chloroquine within 14 days prior to the study vaccination through to Day 28

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety | Day 0-180
  Safety defined as frequency and severity of vaccine-related reactogenicity events and reported AEs
Immunogenicity | Day 0-28
  Immunogenicity as defined as rate of seroconversion (4-fold rise) of serum Inaba vibriocidal antibody and initial estimates of between subject variability of vibriocidal antibody response

SECONDARY OUTCOMES:
Kinetics | Day 0-28
  Kinetics of serum Inaba vibriocidal antibody after 1 oral dose of CVD 103-HgR
Serum anti-cholera toxin (CT) IgG antibody conversion rates | Day 0-28
  Anti-cholera toxin IgG antibody conversion rates
Fecal shedding | Day 0-7
  Fecal shedding of CVD 103-HgR by vaccine recipient
Vibriocidal seroconversion and shedding of CVD 103-HgR in household contacts | Day 0-28
  Vibriocidal seroconversion and shedding of CVD 103-HgR in household contacts

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Derived] Chen WH, Greenberg RN, Pasetti MF, Livio S, Lock M, Gurwith M, Levine MM. Safety and immunogenicity of single-dose live oral cholera vaccine strain CVD 103-HgR, prepared from new master and working cell banks. Clin Vaccine Immunol. 2014 Jan;21(1):66-73. doi: 10.1128/CVI.00601-13. Epub 2013 Oct 30. PMID 24173028
- See also: PubMed (results) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3910924/